CLINICAL TRIAL: NCT02152670
Title: Understanding Dopamine Mechanisms in Cocaine Addiction Using AMPT and Methylphenidate With [11C]RAC/[11C]PHNO PET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study drug became unaffordable for the purposes of the research.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 1403013567
Record Dates: First submitted 2014-05-20; First posted 2014-06-02 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Methylphenidate; alpha-Methyltyrosine; naxagolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Baseline (Experimental): Subjects will receive 2 baseline PET scans with the radioligands (11C)(+)PHNO and (11C)(+)raclopride
  Interventions: Other: [11C]PHNO; Other: [11C]raclopride
- Dopamine Release (Experimental): Subjects will receive 1 PET scan following a PO dose of 60mg of methylphenidate to facilitate dopamine release with the radioligand (11C)(+)PHNO
  Interventions: Drug: Methylphenidate; Other: [11C]PHNO
- Endogenous Dopamine (Experimental): Subjects will receive 2 PET scans following 48 hours of dopamine depletion via AMPT with the radioligands (11C)(+)PHNO and (11C)(+)raclopride
  Interventions: Drug: Alpha Methyl Para Tyrosine (AMPT); Other: [11C]PHNO; Other: [11C]raclopride

INTERVENTIONS:
Drug: Methylphenidate
  Arms: Dopamine Release
Drug: Alpha Methyl Para Tyrosine (AMPT)
  Arms: Endogenous Dopamine
Other: [11C]PHNO
Other: [11C]raclopride
  Arms: Baseline; Endogenous Dopamine

SUMMARY:
Studies using positron emission tomography (PET) have been used with great success in demonstrating specific abnormalities in several facets of dopaminergic system function in human populations (Narendran and Martinez 2009). Among the first, most consistent, and broadly replicated of such findings in drug- (including cocaine) dependent individuals has been the reduction in subcortical (striatal) D2/3 receptors as imaged, most commonly, by the reversible, non-selective, D2/3 receptor antagonist radiotracer, [11C]raclopride. Certain dissociations on D2/3 availability by radioligand ([11C]raclopride vs. [11C]PHNO) and by brain region (striatum vs. SN; terminal vs. somatodendritic, respectively) are poorly understood in relationship to prior antagonist tracer results. In the current study the investigators will use pharmacological interventions (AMPT and methylphenidate) with both antagonist and agonist radiotracers to experimentally reconcile these discordant findings and clarify potential mechanistic inter-relationships.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 50 years,
2. voluntary, written, informed consent,
3. physically healthy by medical history, physical, neurological, ECG, and laboratory examinations,
4. for females, non-lactating, no longer of child-bearing potential (or agree to practice effective contraception during the study), and a negative serum pregnancy (B-HCG) test.
5. English speaking
6. No other major Axis DSM-IV diagnosis present, besides required as below

Inclusion criteria for cocaine dependent:

1. DSM-IV criteria for Cocaine Abuse (305.60) or Cocaine Dependence (304.20)
2. recent street cocaine use,
3. intravenous and/or smoked (crack/ freebase) use,
4. positive urine toxicology screen for cocaine,

Inclusion criteria for healthy controls:

1. No current, or history of, any DSM-IV diagnosis
2. No first-degree relative with history of psychotic, mood, or anxiety disorder

Exclusion Criteria:

1. medical contraindications to AMPT administration (e.g., known sensitivity/reaction to AMPT);
2. medical contraindications to MPH administration (e.g., history of cardiac problems, seizures, etc.)
3. drug or alcohol dependence (except nicotine),
4. a primary major DSM-IV psychiatric diagnosis (schizophrenia, bipolar disorder, etc.), unrelated to cocaine or pathological gambling
5. positive answers on the cardiac screening questionnaire that may place the subject at higher risk, as determined by cardiologist review of both the questionnaire responses and screening ECG
6. current use of psychotropic and/or potentially psychoactive prescription medication,
7. physical or laboratory (B-HCG) evidence of pregnancy,
8. clotting disorders or recent anticoagulant therapy,
9. MRI-incompatible implants and other contraindications for MRI (i.e., aneurysm clip, metal fragments, internal electrical devices such as a cochlear implant, spinal cord stimulator or pacemaker),
10. history of claustrophobia or feeling of inability to lie still on his back for the PET or MRI scans,
11. history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over Radioactive Drug Research Committee (RDRC) limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.
12. donation or loss of 550 mL of blood or more (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to the first dose of study drug.
13. use any prescription medications and/or over-the-counter medications, vitamins and/or herbal supplements within 2 weeks prior to study and for the duration of the study without approval from the study doctor.
14. eat grapefruit or grapefruit products, and drink alcohol, and anything containing caffeine 3 days before study and during study
15. For CD subjects, < 1 year of cocaine dependence, .
16. Subjects with current, past, or anticipated exposure to radiation in the workplace.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06-09 (Actual); Study Completion 2014-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Malison, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled and Randomized: This summarizes the single patient enrolled and randomized to the study.
Period: Overall Study
Arm/Group | Enrolled and Randomized
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only 1 single patient was enrolled and randomized.
Arm/Group | Enrolled and Randomized
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: BPND
Description: BPND is a measure of dopamine receptor availability
Time Frame: 2 weeks
Population: Only a single patient was enrolled and randomized.
Arm/Group | Enrolled and Randomized
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Enrolled and Randomized
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes